CLINICAL TRIAL: NCT03197103
Title: The Impact of N-Acetylcysteine on Volumetric Retention of Autologous Fat Graft for Breast Asymmetry Correction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Bartłomiej Noszczyk, Ph.D., M.D., Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 58/IX/PB/Noszczyk/16
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Breast; Deformity, Congenital; Graft Loss; Adipose Tissue Atrophy; Breast; Atrophy
Keywords: Autologous fat grafting; Breast; Deformity; Asymmetry; Tuberous breast; Acetylcysteine
MeSH Terms: conditions — Congenital Abnormalities; Atrophy | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine (NAC) (Experimental): Breast enlargement with autologous fat graft obtained by liposuction with Pietruski solution (tumescent solution with NAC).
  Interventions: Drug: N-Acetylcysteine (NAC)
- Control (No Intervention): Contralateral breast enlargement with autologous fat graft obtained by liposuction with standard tumescent solution.

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) — For more information read Experimental Arm description
  Other Names: Acetylcysteine
  Arms: N-Acetylcysteine (NAC)

SUMMARY:
The aim of this study is to assess the effect of new tumescent solution for liposuction containing N-Acetylcysteine (Pietruski solution) on the autologous fat graft volumetric retention used for healthy women breast asymmetry correction by means of lipofilling.

DETAILED DESCRIPTION:
Lipofilling is the process of relocating autologous fat to change the volume, shape, and profile of tissues. It is considered a simple, inexpensive and minimally invasive technique indicated for both congenital and acquired soft tissue defects in many sites. Success is heavily dependent on the harvesting technique, preparing and injection of the fat. The main limitation of the abovementioned surgical procedure is a loss of transplanted adipose tissue which is believed to be caused mainly by cells injury in oxidative, ischemic, and mechanical stress mechanism. High graft resorption rate results in undercorrection and requirement for multiple-stage treatment. The aim of this study is to assess the effect of new tumescent solution for liposuction containing N-Acetylcysteine (NAC) on the autologous fat graft volumetric retention used for healthy women breast asymmetry correction by means of lipofilling. NAC reduces free radicals using a sulfhydryl chemical group. In authors opinion, this antioxidant effect may decrease oxidative stress experienced by adipose graft cells during the harvest procedure, therefore potentially improving the long-term survivability of the fat graft, lowering the number of re-operations and even maybe the total volume of fat graft needed to achieve satisfactory results. The results of this study may justify the usage of novel tumescent solution (Pietruski solution) for autologous adipose tissue graft harvest in the routine clinical setting.

The subjects for this project will consist of the group of women who are candidates for hypoplastic, asymmetric breasts correction with at least two-staged lipofilling procedure. The bilateral character of such defect allows for each patient to serve as her own control. In the first lipofilling procedure one breast will be enlarged with autologous fat graft harvested from one thigh region after its infiltration with Pietruski solution. The contralateral breast will be enlarged with adipose tissue collected from contralateral thigh area by performing lipoaspiration after standard tumescent solution infiltration. Only the first stage of breasts defect correction is included in this study. Additional, future lipofilling procedures will utilize fat graft obtained with a standard tumescent solution only.

The hypothesis that addition of NAC to the tumescent solution used for the fat graft harvest procedure will decrease its long-term resorption in breast region will be tested in comparison to the fat graft obtained with liposuction using standard tumescent solution. For each subject, a breast magnetic resonance imaging (MRI) will be performed before and six months after the first fat graft transfer enabling quantitative, volumetric analysis of the transplanted adipose tissue resorption. In addition, a volume of 50 ml of each harvested fat graft will be intended for genetic and immunohistochemical analysis. The results will be compared using two-tailed t-tests with statistical significance set at p<0.05.

The study will be conducted at the Plastic Surgery Department, Centre of Postgraduate Medical Education, Warsaw, Poland.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-40 years
* BMI > 20
* Breasts asymmetry (including tuberous breasts deformity) with indications for treatment with autologous fat grafting
* ASA PS I

Exclusion Criteria:

* Asthma
* A history of allergic reaction to NAC
* Peptic ulcer disease
* Contraindications to MRI imaging
* A history of breast surgery or radiotherapy
* A history of hip/thigh surgery or injury
* Breastfeeding, pregnancy or planned pregnancy within a year
* Ilness or general state of health precluding general anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Autologous fat graft volumetric analysis | 6 months following the intervention in the last enrolled participant
  Volumetric analysis of fat graft six months after operation (postoperative breast adipose tissue volume in comparison to preoperative volume).

SECONDARY OUTCOMES:
Intraoperative complications | During intervention (operation)
  Any complication that occurred during the lipofilling procedure.
Postoperative complications | 6 months following the intervention
  Any complication or adverse effect of the lipofilling procedure that occurred in the six-month time frame following the operation.
Immunohistochemical and genetic analysis of lipoaspirates. | Immediately after intervention
  A volume of at least 50 ml of each harvested fat graft (control tumescent solution vs Pietruski tumescent solution) will be intended for genetic and immunohistochemical analysis. The immediate analysis will include oxidative stress markers quantification (Nitric Oxide, Superoxide dismutase, Reactive Oxygen Species), dead cell count evaluation (flow cytometry) and RNA isolation for the future qRT-PCR analysis of chosen targets expression related to cells' stress response. Additional, an attempt will be taken to isolate adipose-derived stem cells (ASC) from each lipoaspirate for the purpose of hydrogen peroxide exposure test, ELISA test, flow cytometry, Colony Forming Unit-Fibroblastic Assay (CFU-F) and Cell Proliferation Assay.

CONTACTS AND LOCATIONS:
Overall Officials: Bartłomiej Noszczyk, Ph.D., M.D., Study Director — Centre of Postgraduate Medical Education; Piotr Pietruski, M.D., Principal Investigator — Centre of Postgraduate Medical Education
Locations (1):
- Centre of Postgraduate Medical Education, Prof. W. Orlowski Memorial Hospital, Warsaw, Mazowiecki, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pietruski P, Paskal W, Paluch L, Paskal AM, Nitek Z, Wlodarski P, Walecki J, Noszczyk B. The Impact of N-Acetylcysteine on Autologous Fat Graft: First-in-Human Pilot Study. Aesthetic Plast Surg. 2020 May 18. doi: 10.1007/s00266-020-01730-1. Online ahead of print. PMID 32424535
- [Derived] Pietruski P, Paskal W, Paluch L, Paskal AM, Nitek Z, Wlodarski P, Walecki J, Noszczyk B. The Impact of N-Acetylcysteine on Autologous Fat Graft: First-in-Human Pilot Study. Aesthetic Plast Surg. 2021 Oct;45(5):2397-2405. doi: 10.1007/s00266-020-01633-1. Epub 2020 Mar 27. PMID 32221675